

## **SYNOPSIS**

| SYNOPSIS | |
|---|---|
| Protocol No. | BR-FMS-PASS-401 |
| Sponsor | Boryung Pharmaceutical Co., Ltd. |
| Active Ingredient<br>Name | Fimasartan potassium trihydrate |
| Study Title | A Prospective, Observational, Post-Authorization Long-term Safety Surveillance on Antihypertensive Treatment With Kanarb® (Fimasartan) During 1 Year Among 20 and Older Diagnosed With Essential Hypertension |
| Study Objectives | Primary Objective: |
| | To evaluate the incidence and characteristics (profile, relationship to the study drug, severity, and outcome) of adverse events (AEs) observed during 1-year treatment with Kanarb tablet® (fimasartan) |
| | Secondary Objectives: |
| | To investigate the rates of discontinuation and persistence of 1-year treatment with Kanarb tablet <sup>®</sup> (fimasartan) (including the investigation of the rates of switching to other drugs and concomitant administration with other antihypertensive drugs) |
| No. of Subject | Target number of subjects: 600 subjects |
| Inclusion Criteria | 1. Patients with essential hypertension |
| | 2. Taking Kanarb tablet $^{\mathbb{R}}$ (fimasartan) as prescribed previously (within 1 month) or newly |
| | 3. Male and female adults aged 20 years or older |
| | 4. Voluntarily provided a written consent to participate in the study |
| <b>Exclusion Criteria</b> | Meeting any of the following including contraindications for fimasartan |
| | 1. Patients with hypersensitivity to this drug or the ingredients of this drug |
| | 2. Pregnant or breast-feeding women |
| | 3. Patients on renal dialysis |
| | 4. Patients with moderate to severe hepatic impairment |
| | 5. Patients with biliary atresia |
| | 6. Genetic disorders such as galactose intolerance, lapp lactase deficiency, or glucose-galactose malabsorption |
| | 7. Patients considered inappropriate for taking Kanarb tablet® (fimasartan) by investigator |
| | 8. Clinically significant abnormal liver function (AST, ALT ≥2 x upper limit of normal (ULN); TB ≥1.5 ULN) |
| Statistical<br>Analysis Method | Incidence of adverse events (AEs), treatment persistence rate and treatment discontinuation rate of fimasartan were reported for each measurement time point and their 95% confidence intervals were presented |